CLINICAL TRIAL: NCT02599337
Title: Randomized, Open-label, 3-way Reference Replicated Crossover Bioequivalence Study of Sorafenib 200 mg Tablet and Nexavar (Reference) Following a 200 mg Dose in Healthy Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Sorafenib Tablet and Nexavar
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yabao Pharmaceutical Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 150230
Record Dates: First submitted 2015-10-20; First posted 2015-11-06 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-07

CONDITIONS: Fasting
Keywords: bioequivalence
MeSH Terms: conditions — Fasting | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- sorafenib (Experimental): Sorafenib is the test product.In period 1, period 2 and period 3, 12 of 36 Subjects were given Single oral dose (1 x 200 mg) sarofenib.
  Interventions: Drug: Nexavar; Drug: Sorafenib
- Nexavar (Active Comparator): Nexavar is the reference product.In period 1, period 2 and period 3, 24 of 36 Subjects were given Single oral dose (1 x 200 mg) Nexavar .
  Interventions: Drug: Nexavar; Drug: Sorafenib

INTERVENTIONS:
Drug: Nexavar — Single oral dose (1 x 200 mg) sorafenib or Nexavar in each period. No food were allowed from at least 10 hours before dosing until at least 4 hours after dosing.
  Except for water given with study medication, no fluids were allowed from 1 hour before dosing until 1 hour post-dose.
Drug: Sorafenib — Single oral dose (1 x 200 mg) sorafenib or Nexavar in each period. No food were allowed from at least 10 hours before dosing until at least 4 hours after dosing.
  Except for water given with study medication, no fluids were allowed from 1 hour before dosing until 1 hour post-dose.
  Other Names: sarafenib

SUMMARY:
Randomized, open-label, 3-way reference replicated crossover bioequivalence study of sorafenib 200 mg tablet and nexavar (reference) following a 200 mg dose in healthy subjects under fasting conditions.

DETAILED DESCRIPTION:
This will be a single centre, bioequivalence, open-label, randomized, single-dose, 3-period, 3-sequence, reference replicated, crossover study. 36 healthy adult males or non-childbearing potential females, ≥18 and ≤65 years of age, smoker and/or non-smoker.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-childbearing potential female, which includes post-menopausal female (absence of menses for 12 months prior to drug administration, bilateral oophorectomy or hysterectomy with bilateral oophorectomy at least 6 months prior to drug administration) or surgically sterile female (hysterectomy or tubal ligation at least 6 months prior to drug administration), smoker (no more than 25 cigarettes or equivalent daily) or non-smoker, ≥18 and ≤65 years of age, with BMI >18.5 and <30.0 kg/m2 and body weight ≥50.0 kg for males and ≥45.0 kg for females.
2. Healthy as defined by:

   * the absence of clinically significant illness and surgery within 4 weeks prior to dosing. Subjects vomiting within 24 hours pre-dose will be carefully evaluated for upcoming illness/disease. Inclusion pre-dosing is at the discretion of the Qualified Investigator.
   * the absence of clinically significant history of neurological, endocrinal, cardiovascular, pulmonary, hematological, immunologic, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
   * lipase within normal laboratory ranges
3. Capable of consent.

Exclusion Criteria:

1. Any clinically significant abnormality or abnormal laboratory test results found during medical screening or positive test for hepatitis B, hepatitis C, or HIV found during medical screening.
2. Positive urine drug screen at screening.
3. History of allergic reactions to sorafenib, any of the excipients or other related drugs.
4. Use of any drugs known to induce or inhibit CYP3A4 metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, etc.; examples of inhibitors: HIV antivirals, clarithromycin, ciprofloxacin, gestodene, etc. within 30 days prior to the first study drug administration.
5. Positive pregnancy test at screening.
6. Any reason which, in the opinion of the Qualified Investigator, would prevent the subject from participating in the study.
7. Clinically significant electrocardiogram (ECG) abnormalities (QTc >450) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
8. History of significant alcohol abuse within one year prior to screening or regular use of alcohol within six months prior to the screening visit (more than fourteen units of alcohol per week [1 unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]).
9. History of significant drug abuse within one year prior to screening or use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP], and crack) within 1 year prior to screening.
10. Participation in a clinical trial involving the administration of an investigational or marketed drug within 30 days (90 days for biologics) prior to the first dosing or concomitant participation in an investigational study involving no drug administration.
11. Use of medication other than topical products without significant systemic absorption:

    * prescription medication within 14 days prior to the first dosing;
    * over-the-counter products including natural health products (e.g. food supplements and herbal supplements) within 7 days prior to the first dosing, with the exception of the occasional use of acetaminophen (up to 2 g daily);
    * a depot injection or an implant of any drug within 3 months prior to the first dosing.
12. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dosing.
13. Hemoglobin <128 g/L (males) and <115 g/L (females) and hematocrit <0.37 L/L (males) and <0.32 L/L (females) at screening.
14. Breast-feeding subject.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Assessment of the bioequivalence of sorafenib tablet (Test)and Nexavar(Reference), on day 4. | 96 hours
  Compare the rate and extent of absorption of sorafenib 200 mg tablet (Test) versus Nexavar (Reference), administered as 1 x 200 mg tablet under fasting conditions. Evaluate whether has the bioequivalence between the Test and the Reference.Criteria as follows: for a primary parameter (AUC0-t, AUC0-inf, or Cmax), if
  1. the point estimate of the Test-to-Reference ratio must be within 80.00% 125.00%, and
  2. the 95% upper confidence bound for the scaled average bioequivalence criterion must be equal to or less than zero (≤0) to conclude in favor of BE for that parameter.

SECONDARY OUTCOMES:
safety: number TEAEs, deaths, SAEs and other significant adverse events | 96 hours
  Number of Treatment-Emergent Adverse Events(TEAEs). Number of deaths. Number of SAEs. Number of other significant adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Larouche, MD, Principal Investigator — employee
Locations (1):
- Inventiv Health Clinique Inc., Québec, Quebec, Canada